CLINICAL TRIAL: NCT01151891
Title: The Natural History of Pedal Puncture Wounds in Diabetics: a Cross-sectional Survey in the Parish of St. James, Jamaica.
Brief Title: Natural History of Pedal Puncture Wounds in Diabetics
Status: Completed | Type: Observational
Sponsor: Cornwall Regional Hospital (Other Government)
Collaborators: St. James Health Department (Unknown); Private Practice of Dr. Hector Robinson (Unknown); Private Practice of Dr. Curtis Yeates (Unknown)
Responsible Party: Jeffrey East, Cornwall Regional Hospital
Other Study IDs: JE-2
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes
Keywords: Pedal puncture wounds; Infection in pedal puncture wounds; Diabetes education and pedal puncture wounds
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetics: Diabetics in the parish of St. James, Jamaica

SUMMARY:
There are no evidence (research) based guidelines for treatment of early, closed puncture wounds of the feet in diabetics. Surgeons usually see only the limb- and life-threatening consequences of puncture wounds of the feet in diabetics, and are therefore tempted to advocate more aggressive, preemptive, invasive primary treatment for all such wounds, assuming, from this blinkered perspective that all such wounds progress to serious infection. This study is designed to determine the natural history of puncture wounds of the feet in diabetics, specifically, whether all become infected or whether some do heal without any surgical intervention. It requires administration of a questionnaire to 188 known diabetics attending 11 selected outpatient health care centers in the parish of St. James, Jamaica.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic
* 15 years and older
* Resident in the parish of St. James, Jamaica

Exclusion Criteria:

* Impairment of conscious level or mental status such that autonomy is compromised

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetics attending 3 public hospital outpatient clinics, 6 public Health Center primary care clinics and 2 private Internist's clinics.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pedal puncture wounds | September, 2010

SECONDARY OUTCOMES:
Infection in pedal puncture wounds | September, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M East, MD, Principal Investigator — Cornwall Regional Hospital
Locations (4):
- Jamaica (4):
  - Cornwall Regional Hospital, Montego Bay, Saint James Parish
  - Health Centers of the St. James Health Department, Montego Bay, Saint James Parish
  - Private clinic of Dr. Curtis Yeates, Montego Bay, Saint James Parish
  - Private clinic of Dr. Hector Robinson, Montego Bay, Saint James Parish

REFERENCES:
- [Background] Wilks RJ, Sargeant LA, Gulliford MC, Reid ME, Forrester TE. Management of diabetes mellitus in three settings in Jamaica. Rev Panam Salud Publica. 2001 Feb;9(2):65-72. doi: 10.1590/s1020-49892001000200002. PMID 11293831
- [Background] Frykberg RG, Zgonis T, Armstrong DG, Driver VR, Giurini JM, Kravitz SR, Landsman AS, Lavery LA, Moore JC, Schuberth JM, Wukich DK, Andersen C, Vanore JV; American College of Foot and Ankle Surgeons. Diabetic foot disorders. A clinical practice guideline (2006 revision). J Foot Ankle Surg. 2006 Sep-Oct;45(5 Suppl):S1-66. doi: 10.1016/S1067-2516(07)60001-5. PMID 17280936
- [Background] Fitzgerald RH Jr, Cowan JD. Puncture wounds of the foot. Orthop Clin North Am. 1975 Oct;6(4):965-72. PMID 241038
- [Background] Joseph WS, LeFrock JL. Infections complicating puncture wounds of the foot. J Foot Surg. 1987 Jan-Feb;26(1 Suppl):S30-3. PMID 2881957
- [Background] Verdile VP, Freed HA, Gerard J. Puncture wounds to the foot. J Emerg Med. 1989 Mar-Apr;7(2):193-9. doi: 10.1016/0736-4679(89)90269-2. PMID 2567749
- [Background] Weber EJ. Plantar puncture wounds: a survey to determine the incidence of infection. J Accid Emerg Med. 1996 Jul;13(4):274-7. doi: 10.1136/emj.13.4.274. PMID 8832349
- [Background] Lavery LA, Armstrong DG, Wunderlich RP, Mohler MJ, Wendel CS, Lipsky BA. Risk factors for foot infections in individuals with diabetes. Diabetes Care. 2006 Jun;29(6):1288-93. doi: 10.2337/dc05-2425. PMID 16732010
- [Background] Wright-Pascoe R, Roye-Green K, Bodonaik N. The medical management of diabetes mellitus with particular reference to the lower extremity: the Jamaican experience. West Indian Med J. 2001 Mar 1-4;50 Suppl 1:46-9. PMID 15973818
- [Derived] East JM, Yeates CB, Robinson HP. The natural history of pedal puncture wounds in diabetics: a cross-sectional survey. BMC Surg. 2011 Oct 17;11:27. doi: 10.1186/1471-2482-11-27. PMID 22004373